CLINICAL TRIAL: NCT00612482
Title: Youth Substance Use Prevention/Reduction Through Science-based Drug Abuse Education: A High School Pilot Study
Brief Title: Youth Substance Use Prevention/Reduction Through Science-based Drug Abuse Education
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Boston Public Schools (Other)
Responsible Party: Sion Kim Harris, Children's Hospital Boston
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 06120537
Record Dates: First submitted 2008-01-29; First posted 2008-02-11 (Estimated); Last update posted 2011-03-14 (Estimated); Status verified 2011-03

CONDITIONS: Substance Abuse
Keywords: Substance abuse
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention): Participants in the "no intervention" condition will receive the usual high school science curriculum.
- 2 (Experimental): Participants in the "experimental" arm will receive the 5-lesson, science-based substance abuse prevention curriculum in their science classes.
  Interventions: Other: drug prevention curriculum

INTERVENTIONS:
Other: drug prevention curriculum — Participants in the "experimental" arm of the study will receive the 5-lesson, science-based drug prevention curriculum in their science classes.
  Arms: 2

SUMMARY:
Our primary goal is to conduct a pilot study of the effects of a new potential strategy for youth substance abuse prevention - science-based drug education integrated into the high school science curriculum. Through this pilot study we propose to: (1) demonstrate that this new strategy shows promise, and (2) estimate the effect size for the intervention.

DETAILED DESCRIPTION:
NIDA, in recent years, has put resources into summarizing and synthesizing cutting-edge medical and basic science research discoveries about the short-term and long-term effects of drug use on the developing brain. One outcome of this results was the production of a science-based drug education program entitled "The Brain: Understanding Neurobiology Through the Study of Addiction." This is a 5-lesson module for high school science classes that teaches about brain structure and function, how drugs affect and change the biology and chemistry of the brain, how addiction occurs in the brain, and that addiction is a chronic, recurring disease. However, the effect of receipt of this program on students' substance use knowledge, attitudes, perceived risk of harm, and behavior has not been systematically evaluated to date.

The specific aims of this project are:

1. To evaluate the effects of receipt of the curriculum on specific cognitive contributors to substance use including a)students' knowledge about the short- and long-term effects of substance use on the brain; b)perceived risk of harm from substance use; and c)intention to use substances in the next 3 months.
2. To evaluate the effects of the intervention on actual substance use behavior. We hypothesize that the effectiveness of this approach may be modified by the students' level of prior and current substance use, with the effect being stronger among those who have not already initiated use, or among those who have very low use. Therefore, we will specifically examine whether the intervention a)prevents substance use initiation among students who had no previous use, b)stops use among students with low lifetime use, and c) reduces use among those with higher levels of use.

ELIGIBILITY:
Inclusion Criteria:

* Student in 9th/10th/11th grade science classes at Fenway High School at start of study or student in 11th grade science classes at Boston Arts Academy at start of study
* Parental permission to participate

Exclusion Criteria:

* No parental permission to participate
* Unable to read English

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 225 (Actual)
Dates: Start 2006-12; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Lifetime, past 6 month and past 30 day use of substances | Pre-intervention, immediate post-intervention, 6-7 month post-intervention

SECONDARY OUTCOMES:
Frequency and quantity of substance use | Pre-intervention, immediate post-intervention, 6-7 months post-intervention
Knowledge about effects of substance use on the brain | Pre-intervention, immediate post-intervention, 6-7 months post-intervention
Perceived risk of harm of substance use | Pre-intervention, immediate post-intervention, 6-7 months post-intervention
Intention to use substances in the next 3 months | Pre-intervention, immediate post-intervention, 6-7 months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Sion Kim Harris, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

REFERENCES:
- See also: Web page of the Center for Adolescent Substance Abuse Research — http://www.ceasar.org